CLINICAL TRIAL: NCT06240260
Title: Utilization of Transcutaneous Electrical Nerve Stimulation (TENS) Unit for Analgesia During IUD Insertion: A Prospective Cohort Study
Brief Title: TENS Unit for Analgesia During IUD Insertion
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY00004077
Record Dates: First submitted 2023-11-27; First posted 2024-02-05 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: IUD; Analgesia; Patient Preference; Pain, Acute
Keywords: iud; contraception; iud placement; pain management; teen
MeSH Terms: conditions — Agnosia; Patient Preference; Acute Pain; Stillbirth | interventions — Transcutaneous Electric Nerve Stimulation; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- TENS unit (Experimental): Patients who choose to use a TENS unit for their IUD insertion procedure
  Interventions: Device: TENS (transcutaneous electrical nerve stimulation) unit
- Standard care (Active Comparator): Patients who decline to use a TENS unit for their IUD insertion procedure
  Interventions: Other: Standard care

INTERVENTIONS:
Device: TENS (transcutaneous electrical nerve stimulation) unit — Transcutaneous electrical nerve stimulation (TENS) is a method of pain relief involving the use of a mild electrical current.
  A TENS machine is a small, battery-operated device that has leads connected to sticky pads called electrodes.
  Other Names: TENS (transcutaneous electrical nerve stimulation) machine
  Arms: TENS unit
Other: Standard care — Paracervical block only or participant declines analgesia for IUD insertion
  Arms: Standard care

SUMMARY:
Subjects will be screened over the phone or in Tufts GYN clinic for participation in the study. If eligible and interested in participating, written informed consent (and assent if applicable) will be obtained. After informed consent/assent, the patient will be enrolled in the study. The patient will decide if they desire to use TENS unit during IUD insertion appointment and inform the study team. The clinic visit will proceed as normal, with additional study proceedings as follows. The study personnel will complete the 'Background Questionnaire' with the patient prior to IUD insertion. During the IUD insertion appointment, study personnel will assist in collection of the 'Study visit' data collection form. This includes recording the patient's pain score at various time points throughout the insertion procedure:

* anticipated pain during IUD insertion
* baseline pain prior to insertion
* speculum insertion
* tenaculum placement
* paracervical block administration (if performed)
* cervical dilation (if performed)
* uterine sounding
* IUD insertion
* 5 minutes after IUD insertion

Study personnel will also time the insertion procedure and collect additional data as outlined in the 'Study visit data collection form.' After IUD insertion, the participant will be asked to complete the 'Post-IUD Insertion Survey.' Once this survey is complete, this will conclude the study participation. Participation will last through the study visit only.

As part of the standard of care, a urine pregnancy test will be obtained and confirmed negative prior to IUD insertion. Patients will receive routine pain management modalities per shared decision-making with their clinical provider which may include NSAID administration, paracervical block, and heating pad.

ELIGIBILITY:
Inclusion Criteria:

1. Persons with a uterus desiring insertion of intrauterine device
2. Able to provide informed consent/assent
3. Age 12-50 years old
4. Minors 12 years of age and older will be included in the study if postmenarchal

Exclusion Criteria:

1. Unable to provide informed consent/assent
2. Prior cervical procedure (ie loop electrosurgical excision procedure, LEEP)
3. Concurrent cervical or intrauterine procedure (ie colposcopy or dilation and curettage)
4. Cutaneous damage at the TENS electrode sites
5. Chronic or pre-procedure use of opioids
6. Chronic pain diagnosis
7. Prior IUD insertion
8. Any contraindication to intrauterine device (IUD):

   1. Pregnancy
   2. Uterine anomaly that distorts the uterine cavity
   3. Acute pelvic inflammatory disease (PID)
   4. Postpartum endometritis or infected abortion in the past 3 months
   5. Unexplained abnormal uterine bleeding
   6. Wilson's disease or copper allergy (contraindication to copper IUD only)
   7. Breast cancer (contraindication to levonorgestrel IUD only

Ages: 12 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-04-30 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Self reported pain intensity from participants during IUD insertion | Day 1
  Survey responses

SECONDARY OUTCOMES:
Pain at other time points during IUD insertion procedure | Day 1
  Survey responses
Rate of vasovagal responses | Day 1
  Participant observation
Likelihood to recommend pain management regiment to a friend for same procedure | Day 1
  Survey responses

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Zuckerman, MD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Seyss R. [Bone scan of persisting epiphyseal cartilage]. Fortschr Geb Rontgenstr Nuklearmed. 1974 Nov;121(5):655-6. No abstract available. German. PMID 4141332
- [Background] Asker C, Stokes-Lampard H, Beavan J, Wilson S. What is it about intrauterine devices that women find unacceptable? Factors that make women non-users: a qualitative study. J Fam Plann Reprod Health Care. 2006 Apr;32(2):89-94. doi: 10.1783/147118906776276170. PMID 16824298
- [Background] Hurwitz S. Pigmented nevi. Semin Dermatol. 1988 Mar;7(1):17-25. No abstract available. PMID 3153421
- [Background] Kavanaugh ML, Frohwirth L, Jerman J, Popkin R, Ethier K. Long-acting reversible contraception for adolescents and young adults: patient and provider perspectives. J Pediatr Adolesc Gynecol. 2013 Apr;26(2):86-95. doi: 10.1016/j.jpag.2012.10.006. Epub 2012 Dec 31. PMID 23287602
- [Background] Callahan DG, Garabedian LF, Harney KF, DiVasta AD. Will it Hurt? The Intrauterine Device Insertion Experience and Long-Term Acceptability Among Adolescents and Young Women. J Pediatr Adolesc Gynecol. 2019 Dec;32(6):615-621. doi: 10.1016/j.jpag.2019.08.004. Epub 2019 Aug 8. PMID 31401254
- [Background] ACOG Committee Opinion No. 735: Adolescents and Long-Acting Reversible Contraception: Implants and Intrauterine Devices. Obstet Gynecol. 2018 May;131(5):e130-e139. doi: 10.1097/AOG.0000000000002632. PMID 29683910
- [Background] American College of Obstetricians and Gynecologists' Committee on Gynecologic Practice; Long-Acting Reversible Contraceptive Expert Work Group. Committee Opinion No 672: Clinical Challenges of Long-Acting Reversible Contraceptive Methods. Obstet Gynecol. 2016 Sep;128(3):e69-77. doi: 10.1097/AOG.0000000000001644. PMID 27548557
- [Background] Crawford M, Davy S, Book N, Elliott JO, Arora A. Oral Ketorolac for Pain Relief During Intrauterine Device Insertion: A Double-Blinded Randomized Controlled Trial. J Obstet Gynaecol Can. 2017 Dec;39(12):1143-1149. doi: 10.1016/j.jogc.2017.05.014. Epub 2017 Aug 18. PMID 28826645
- [Background] Nagatomo T, Tajiri A, Nakamura T, Hokibara R, Tanaka Y, Aono J, Tsuchihashi H. Adrenergic and serotonergic receptor-blocking potencies of terazosin, a new antihypertensive agent, as assessed by radioligand binding assay. Chem Pharm Bull (Tokyo). 1987 Apr;35(4):1629-32. doi: 10.1248/cpb.35.1629. No abstract available. PMID 2888542
- [Background] Mody SK, Kiley J, Rademaker A, Gawron L, Stika C, Hammond C. Pain control for intrauterine device insertion: a randomized trial of 1% lidocaine paracervical block. Contraception. 2012 Dec;86(6):704-9. doi: 10.1016/j.contraception.2012.06.004. Epub 2012 Jul 6. PMID 22770792
- [Background] Sluka KA, Walsh D. Transcutaneous electrical nerve stimulation: basic science mechanisms and clinical effectiveness. J Pain. 2003 Apr;4(3):109-21. doi: 10.1054/jpai.2003.434. PMID 14622708
- [Background] Rignon-Bret JM, Pompignoli M. [Esthetic presentation]. Inf Dent. 1987 Sep 24;69(32):2757-72. No abstract available. French. PMID 3327829
- [Background] Lison JF, Amer-Cuenca JJ, Piquer-Marti S, Benavent-Caballer V, Bivia-Roig G, Marin-Buck A. Transcutaneous Nerve Stimulation for Pain Relief During Office Hysteroscopy: A Randomized Controlled Trial. Obstet Gynecol. 2017 Feb;129(2):363-370. doi: 10.1097/AOG.0000000000001842. PMID 28079781